CLINICAL TRIAL: NCT05649072
Title: Identifying Underserved Individuals inTexas With Hereditary Cancer Risk Using Mobile Mammography Units and Telegenetics.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Community Outreach and Engagement Fund for Underserved Texans (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-0329; NCI-2022-10036 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Breast Cancer; Colorectal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Colorectal Neoplasms | interventions — Genetic Testing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetic Testing and Counseling (Other): Participants will be given a saliva collection kit to collect a saliva sample for hereditary cancer and genetic testing. The kit includes all standard paperwork and instructions for collecting the sample and shipping the kit back to the genetic testing company (Invitae).
  Interventions: Behavioral: Genetic Testing and Counseling
- Screening Form (Other): Participants will complete a screening form to assess your risk of hereditary breast and colorectal cancers.
  Interventions: Behavioral: Screening Form

INTERVENTIONS:
Behavioral: Genetic Testing and Counseling — Participants will be asked to collect a saliva sample for hereditary cancer and genetic testing
  Arms: Genetic Testing and Counseling
Behavioral: Screening Form — Participant will be answering demographic details
  Arms: Screening Form

SUMMARY:
Identifying women at risk for hereditary cancer potentiates prevention, early detection or personalised treatment against cancer. We using mobile mammography units will provide genetic sceening and testing services to underserved women coming for thier mammograms to these units.

DETAILED DESCRIPTION:
Objectives:

1. To identify underserved women at risk for hereditary breast and colorectal cancers and would be eligible for standard of care genetic counseling and testing using national screening guidelines.
2. To provide education to providers and patients regarding hereditary cancers using previously IRB approved educational material and short video.

ELIGIBILITY:
Inclusion Criteria:

Any woman scheduled at Project VALET mammography screening mobile units will be eligible for this study.

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To identify underserved women at risk for hereditary breast and colorectal cancers eligible for standard-of-care genetic counseling using national screening guidelines. | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Banu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org